CLINICAL TRIAL: NCT02502110
Title: The Study of Rosuvastatin for Reduction of Postoperative Paroxysmal Atrial Fibrillation in Patient Undergoing Radiofrequency Catheter Ablation
Brief Title: Study of Statin for Reduction of Postoperative Paroxysmal Atrial Fibrillation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISSCRES0175
Record Dates: First submitted 2015-07-16; First posted 2015-07-20 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: Atrial Fibrillation; statin; radiofrequency ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rosuvastatin 20mg/day (Experimental): To receive oral rosuvastatin 20mg/day and regular therapy from 7 days before ablation and last for 3 months.
  Interventions: Drug: rosuvastatin
- blank control (No Intervention): Regular therapy from 7 days before ablation and last for 3 months. Regular medicines used for AF includes warfarin, metoprolol sustained release tablet, amiodarone, perindopril and irbesartan.

INTERVENTIONS:
Drug: rosuvastatin — All recruited patients with paroxysmal atrial fibrillation will be randomly allocated to receive oral rosuvastatin 20mg/day or blank control from 7 days before ablation and last for 3 months.
  Other Names: crestor
  Arms: rosuvastatin 20mg/day

SUMMARY:
The study will select all recruited patients with paroxysmal atrial fibrillation will be randomly allocated to receive oral rosuvastatin 20mg/day or blank control from 7 days before ablation and last for 3 months. To observe the early relapse of atrial fibrillation and the changes of white blood cell count, hs-C reactive protein (CRP), interleukin (IL)-6 and tumor necrosis factor (TNF)-α, and the changes of safety indicators .

This study assumes that the early atrial fibrillation (AF) recurrence will be decreased in patients with paroxysmal AF if rosuvastatin 20mg/d is received from 7 days before surgery in these patients who plan to undergo radiofrequency catheter ablation for consecutive 3 months.

DETAILED DESCRIPTION:
This study is a randomized, open-label, multi-centers, parallel-control study to explore whether rosuvastatin 20mg/d could decrease early AF recurrence in patients with paroxysmal AF after radiofrequency catheter ablation. 346 patients with paroxysmal AF are planned to be enrolled. The patients are randomized to receive oral rosuvastatin 20mg/d or control therapy from 7 days before operation and last for 3 months. The early AF recurrence within 90 days after ablation and the changes of 4 inflammatory markers including white blood cell count, hs-CRP, IL-6 and TNF-α and safety indicators will be observed. The study is aim to evaluate the efficacy and safety of rosuvastatin on decreasing early recurrence in patients with paroxysmal AF and discuss its mechanisms of action.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures;
2. Age from 18 to 75 years old, male or female;
3. The course of paroxysmal AF is more than 3 months and confirmed by ECG;
4. Plan to undergo radiofrequency catheter ablation

Exclusion Criteria:

1. Concomitant with serious organic heart disease such as valvular heart diseases, congenital heart diseases, hypertrophic obstructive cardiomyopathy, acute myocardial infarction and unstable angina pectoris;
2. Concomitant with sinoatrial node functional disorder and (or) atrioventricular block;
3. Acute cerebral apoplexy or contraindication of anticoagulant;
4. Thyroid function abnormality;
5. Accepted radiofrequency catheter ablation (RFCA) previously;
6. Being receiving other statins;
7. Be allergic to statins;
8. Pregnancy or women during lactation period;
9. Be not aligning to treatment or follow-up due to mental disorders or other reasons;
10. Be with myopathy or active hepatopathy including agnogenic persistent elevation of serum transaminase and any serum transaminase being over 3 times of upper limit of normal;
11. Be with serious renal dysfunction (creatinine≥3 mg/dL);
12. Need steroid or non-steroid anti-inflammatory drugs to treat inflammation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346 (Estimated)
Dates: Start 2015-08; Primary Completion 2019-03 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
the AF recurrence rate | within 90 days after radiofrequency catheter ablation.

SECONDARY OUTCOMES:
the AF recurrence rate | at 24 hours, 72 hours, 1month, 2 months and 3 months after operation
The inflammatory markers (white blood cell count) | at 24 hours, 72 hours, and 3 months after operation
The inflammatory markers (hs-CRP) | at 24 hours, 72 hours, and 3 months after operation
The inflammatory markers (IL-6) | at 24 hours, 72 hours, and 3 months after operation
The inflammatory markers (TNF-α) | at 24 hours, 72 hours, and 3 months after operation

CONTACTS AND LOCATIONS:
Overall Officials: zhihui zhang, ViceDirector, Principal Investigator — The Third Xiangya Hospital of Central South University

REFERENCES:
- [Background] European Heart Rhythm Association; European Association for Cardio-Thoracic Surgery; Camm AJ, Kirchhof P, Lip GY, Schotten U, Savelieva I, Ernst S, Van Gelder IC, Al-Attar N, Hindricks G, Prendergast B, Heidbuchel H, Alfieri O, Angelini A, Atar D, Colonna P, De Caterina R, De Sutter J, Goette A, Gorenek B, Heldal M, Hohloser SH, Kolh P, Le Heuzey JY, Ponikowski P, Rutten FH. Guidelines for the management of atrial fibrillation: the Task Force for the Management of Atrial Fibrillation of the European Society of Cardiology (ESC). Eur Heart J. 2010 Oct;31(19):2369-429. doi: 10.1093/eurheartj/ehq278. Epub 2010 Aug 29. No abstract available. PMID 20802247
- [Background] Neuman RB, Bloom HL, Shukrullah I, Darrow LA, Kleinbaum D, Jones DP, Dudley SC Jr. Oxidative stress markers are associated with persistent atrial fibrillation. Clin Chem. 2007 Sep;53(9):1652-7. doi: 10.1373/clinchem.2006.083923. Epub 2007 Jun 28. PMID 17599958
- [Background] Anselmi A, Possati G, Gaudino M. Postoperative inflammatory reaction and atrial fibrillation: simple correlation or causation? Ann Thorac Surg. 2009 Jul;88(1):326-33. doi: 10.1016/j.athoracsur.2009.01.031. PMID 19559266
- [Background] Ramlawi B, Otu H, Mieno S, Boodhwani M, Sodha NR, Clements RT, Bianchi C, Sellke FW. Oxidative stress and atrial fibrillation after cardiac surgery: a case-control study. Ann Thorac Surg. 2007 Oct;84(4):1166-72; discussion 1172-3. doi: 10.1016/j.athoracsur.2007.04.126. PMID 17888965
- [Background] Korantzopoulos P, Kolettis T, Siogas K, Goudevenos J. Atrial fibrillation and electrical remodeling: the potential role of inflammation and oxidative stress. Med Sci Monit. 2003 Sep;9(9):RA225-9. PMID 12960937
- [Background] Chimenti C, Russo MA, Carpi A, Frustaci A. Histological substrate of human atrial fibrillation. Biomed Pharmacother. 2010 Mar;64(3):177-83. doi: 10.1016/j.biopha.2009.09.017. Epub 2009 Nov 18. PMID 20006465
- [Background] Kottkamp H, Tanner H, Kobza R, Schirdewahn P, Dorszewski A, Gerds-Li JH, Carbucicchio C, Piorkowski C, Hindricks G. Time courses and quantitative analysis of atrial fibrillation episode number and duration after circular plus linear left atrial lesions: trigger elimination or substrate modification: early or delayed cure? J Am Coll Cardiol. 2004 Aug 18;44(4):869-77. doi: 10.1016/j.jacc.2004.04.049. PMID 15312874
- [Background] Lee SH, Tai CT, Hsieh MH, Tsai CF, Lin YK, Tsao HM, Yu WC, Huang JL, Ueng KC, Cheng JJ, Ding YA, Chen SA. Predictors of early and late recurrence of atrial fibrillation after catheter ablation of paroxysmal atrial fibrillation. J Interv Card Electrophysiol. 2004 Jun;10(3):221-6. doi: 10.1023/B:JICE.0000026915.02503.92. PMID 15133358
- [Background] Sawhney N, Anousheh R, Chen W, Feld GK. Circumferential pulmonary vein ablation with additional linear ablation results in an increased incidence of left atrial flutter compared with segmental pulmonary vein isolation as an initial approach to ablation of paroxysmal atrial fibrillation. Circ Arrhythm Electrophysiol. 2010 Jun;3(3):243-8. doi: 10.1161/CIRCEP.109.924878. Epub 2010 Mar 25. PMID 20339034
- [Background] McCabe JM, Smith LM, Tseng ZH, Badhwar N, Lee BK, Lee RJ, Scheinman MM, Olgin JE, Marcus GM. Protracted CRP elevation after atrial fibrillation ablation. Pacing Clin Electrophysiol. 2008 Sep;31(9):1146-51. doi: 10.1111/j.1540-8159.2008.01155.x. PMID 18834466
- [Background] Kothe H, Dalhoff K, Rupp J, Muller A, Kreuzer J, Maass M, Katus HA. Hydroxymethylglutaryl coenzyme A reductase inhibitors modify the inflammatory response of human macrophages and endothelial cells infected with Chlamydia pneumoniae. Circulation. 2000 Apr 18;101(15):1760-3. doi: 10.1161/01.cir.101.15.1760. PMID 10769273
- [Background] Engelmann MD, Svendsen JH. Inflammation in the genesis and perpetuation of atrial fibrillation. Eur Heart J. 2005 Oct;26(20):2083-92. doi: 10.1093/eurheartj/ehi350. Epub 2005 Jun 23. PMID 15975993
- [Background] Hayashidani S, Tsutsui H, Shiomi T, Suematsu N, Kinugawa S, Ide T, Wen J, Takeshita A. Fluvastatin, a 3-hydroxy-3-methylglutaryl coenzyme a reductase inhibitor, attenuates left ventricular remodeling and failure after experimental myocardial infarction. Circulation. 2002 Feb 19;105(7):868-73. doi: 10.1161/hc0702.104164. PMID 11854129
- [Background] Young-Xu Y, Jabbour S, Goldberg R, Blatt CM, Graboys T, Bilchik B, Ravid S. Usefulness of statin drugs in protecting against atrial fibrillation in patients with coronary artery disease. Am J Cardiol. 2003 Dec 15;92(12):1379-83. doi: 10.1016/j.amjcard.2003.08.040. PMID 14675569
- [Background] Kourliouros A, Valencia O, Hosseini MT, Mayr M, Sarsam M, Camm J, Jahangiri M. Preoperative high-dose atorvastatin for prevention of atrial fibrillation after cardiac surgery: a randomized controlled trial. J Thorac Cardiovasc Surg. 2011 Jan;141(1):244-8. doi: 10.1016/j.jtcvs.2010.06.006. Epub 2010 Jul 10. PMID 20624624
- [Background] Ozaydin M, Varol E, Aslan SM, Kucuktepe Z, Dogan A, Ozturk M, Altinbas A. Effect of atorvastatin on the recurrence rates of atrial fibrillation after electrical cardioversion. Am J Cardiol. 2006 May 15;97(10):1490-3. doi: 10.1016/j.amjcard.2005.11.082. Epub 2006 Mar 29. PMID 16679090
- [Background] Siu CW, Lau CP, Tse HF. Prevention of atrial fibrillation recurrence by statin therapy in patients with lone atrial fibrillation after successful cardioversion. Am J Cardiol. 2003 Dec 1;92(11):1343-5. doi: 10.1016/j.amjcard.2003.08.023. PMID 14636918
- [Background] Almroth H, Hoglund N, Boman K, Englund A, Jensen S, Kjellman B, Tornvall P, Rosenqvist M. Atorvastatin and persistent atrial fibrillation following cardioversion: a randomized placebo-controlled multicentre study. Eur Heart J. 2009 Apr;30(7):827-33. doi: 10.1093/eurheartj/ehp006. Epub 2009 Feb 6. PMID 19202157
- [Background] Patti G, Chello M, Candura D, Pasceri V, D'Ambrosio A, Covino E, Di Sciascio G. Randomized trial of atorvastatin for reduction of postoperative atrial fibrillation in patients undergoing cardiac surgery: results of the ARMYDA-3 (Atorvastatin for Reduction of MYocardial Dysrhythmia After cardiac surgery) study. Circulation. 2006 Oct 3;114(14):1455-61. doi: 10.1161/CIRCULATIONAHA.106.621763. Epub 2006 Sep 25. PMID 17000910
- [Background] Maggioni AP, Fabbri G, Lucci D, Marchioli R, Franzosi MG, Latini R, Nicolosi GL, Porcu M, Cosmi F, Stefanelli S, Tognoni G, Tavazzi L; GISSI-HF Investigators. Effects of rosuvastatin on atrial fibrillation occurrence: ancillary results of the GISSI-HF trial. Eur Heart J. 2009 Oct;30(19):2327-36. doi: 10.1093/eurheartj/ehp357. Epub 2009 Aug 30. PMID 19717850